CLINICAL TRIAL: NCT02449356
Title: Clinical Study of the Endotracheal Tube Used in Prone Position Ventilation Condition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wangyuan Zou (Other)
Collaborators: Central South University (Other)
Responsible Party: Sponsor-Investigator, Wangyuan Zou, postgraduate tutor, Central South University
Organization: Central South University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2013L14
Record Dates: First submitted 2015-04-26; First posted 2015-05-20 (Estimated); Results first posted 2017-06-15 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-03

CONDITIONS: Mechanical Ventilation Complication
Keywords: Prone position ventilation; Endotracheal intubation; Displacement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- prone position endotracheal tube(PPT) (Experimental): the subjects of this arm are given the prone ventilation endotracheal tube which contains fixed device, fixed rope.
  Interventions: Device: prone position endotracheal tube(PPT)
- traditional endotracheal tube(TT) (No Intervention): the subjects of this arm are given the routine endotracheal tube.

INTERVENTIONS:
Device: prone position endotracheal tube(PPT) — some special kind of endotracheal tube,including traditional air tube ,fixed device, fixed rope, and two through holes
  Arms: prone position endotracheal tube(PPT)

SUMMARY:
In this study, the investigators adopt the special endotracheal tube to those patients at prone posture during the operation,or those with acute respiratory distress syndrome in the intensive care unit(ICU), so that the investigators can reduce, or even avoid some severe complications during perianesthesia, and that the investigators can provide strong safeguard measures for the respiratory therapy of critical patients in ICU.

DETAILED DESCRIPTION:
The investigators apply some technical proposals to make it come true:one kind of special endotracheal tube, including traditional endotracheal tube,fixed device,fixed rope,two through holes.With this tube ,the investigators can keep away shifting and falling off of traditional air tube,so that the investigators can try to avoid disaster events.And for the patients with acute respiratory disease syndrome(ARDS),they are always given ventilation in prone position,so it may be beneficial.

ELIGIBILITY:
Inclusion Criteria:

- those who are about to undergo the surgery at prone posture,especially in neurosurgery and spine surgery，American society of anesthesia(ASA) grade I-II，aged from 18 to 65 years old,weight ranged from 50 to 75 kilograms.

Exclusion Criteria:

* No meeting inclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wangyuan Zou, MD,phD, Principal Investigator — Xiangya Hospital
Locations (1):
- Wangyuan Zou, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edgcombe H, Carter K, Yarrow S. Anaesthesia in the prone position. Br J Anaesth. 2008 Feb;100(2):165-83. doi: 10.1093/bja/aem380. PMID 18211991
- [Background] Korn S, Schubert A, Barnett G. Endotracheal tube obstruction during stereotactic craniotomy. J Neurosurg Anesthesiol. 1993 Oct;5(4):272-5. doi: 10.1097/00008506-199310000-00008. PMID 8251716
- [Background] Choi RM, Yoon JS, Noh JH, Kang KO, Ryu SW, Jun HJ, Cho SS. Airway obstruction by extrinsic tracheal compression during spinal surgery under prone position -A case report-. Korean J Anesthesiol. 2010 Dec;59 Suppl(Suppl):S45-8. doi: 10.4097/kjae.2010.59.S.S45. Epub 2010 Dec 31. PMID 21286458
- [Background] Soundararajan N, Cunliffe M. Anaesthesia for spinal surgery in children. Br J Anaesth. 2007 Jul;99(1):86-94. doi: 10.1093/bja/aem120. Epub 2007 May 17. PMID 17510044
- [Background] Tiruvoipati R, Bangash M, Manktelow B, Peek GJ. Efficacy of prone ventilation in adult patients with acute respiratory failure: a meta-analysis. J Crit Care. 2008 Mar;23(1):101-10. doi: 10.1016/j.jcrc.2007.09.003. PMID 18359427
- [Background] Gattinoni L, Carlesso E, Taccone P, Polli F, Guerin C, Mancebo J. Prone positioning improves survival in severe ARDS: a pathophysiologic review and individual patient meta-analysis. Minerva Anestesiol. 2010 Jun;76(6):448-54. PMID 20473258
- [Background] Sud S, Friedrich JO, Taccone P, Polli F, Adhikari NK, Latini R, Pesenti A, Guerin C, Mancebo J, Curley MA, Fernandez R, Chan MC, Beuret P, Voggenreiter G, Sud M, Tognoni G, Gattinoni L. Prone ventilation reduces mortality in patients with acute respiratory failure and severe hypoxemia: systematic review and meta-analysis. Intensive Care Med. 2010 Apr;36(4):585-99. doi: 10.1007/s00134-009-1748-1. Epub 2010 Feb 4. PMID 20130832
- [Background] Zou W, Zhang W, Li X, Guo Q. A randomized crossover comparison of the prone ventilation endotracheal tube versus the traditional endotracheal tube in pediatric patients undergoing prone position surgery. Paediatr Anaesth. 2013 Jan;23(1):98-100. doi: 10.1111/pan.12068. No abstract available. PMID 23216936
- [Derived] Zou W, Shao J, Liang X, Li L, He Z, Guo Q. A randomized comparison of the prone ventilation endotracheal tube versus the traditional endotracheal tube in adult patients undergoing prone position surgery. Sci Rep. 2017 May 11;7(1):1769. doi: 10.1038/s41598-017-02006-6. PMID 28496141

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We have 80 adult patients as candidates who were undergoing the neurosurgery or spinal surgery in Xiangya Hospital affiliated to Central South University between Mar 11, 2014 and Mar 16, 2016. These participants were graded American society of anesthesia(ASA)I-II,and aged 30-70 years old,weighted ranging from 50 to 75 kilograms.
Pre-assignment Details: We finally enrolled 60 patients for our trail. Among the 80 candidates, 7 patients couldn't meet our inclusion criteria; the other 13 patients refused to participate in this trail at last.
Groups:
- Prone Position Endotracheal Tube(PPT): the subjects of this arm are given the prone ventilation endotracheal tube which contains fixed device, fixed rope.
  prone ventilation endotracheal tube: some special kind of endotracheal tube,including traditional air tube ,fixed device, fixed rope, and two through holes
Period: Overall Study
Arm/Group | Traditional Endotracheal Tube(TT) | Prone Position Endotracheal Tube(PPT)
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: all participants in both groups were analyzed
Groups:
- Prone Position Endotracheal Tube(PPT): We enrolled total 60 adult patients undergoing prone position ventilation surgery,and randomized to each group.30 subjects were involved in the prone position endotracheal tube group(PPT), in which group the patients were intubated with the custom-designed endotracheal tube.
- Traditional Endotracheal Tube(TT): We enrolled total 60 adult patients undergoing prone position ventilation surgery,and randomized to each group.30 subjects were involved in the traditional endotracheal tube group(TT), in which group the patients were intubated with the routine endotracheal tube.
- Total: Total of all reporting groups
Arm/Group | Prone Position Endotracheal Tube(PPT) | Traditional Endotracheal Tube(TT) | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: yr] | 49 (5) | 47 (6) | 48 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 15 | 16 | 31
Region of Enrollment [Number; unit: participants]
  China | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Displacement of the Endotracheal Tube
Description: We divided the degree of the displacement of the endotracheal tube into 3 kinds, which included mild(displacement distance<0.5cm),moderate(0.5cm≤displacement distance<1.5cm),severe (1.5cm≤displacement distance).
Time Frame: Participants were followed for the duration of surgery, an average of 2 hours.
Population: All patients in each group were analyzed
Measure: Count of Participants; unit: Participants
Groups:
- Prone Ventilation Endotracheal Tube: the subjects of this arm are given the prone ventilation endotracheal tube which contains fixed device, fixed rope.
  prone ventilation endotracheal tube: some special kind of endotracheal tube,including traditional air tube ,fixed device, fixed rope, and two through holes
- the Traditional Endotracheal Tube: the subjects of this arm are given the routine endotracheal tube.
Arm/Group | Prone Ventilation Endotracheal Tube | the Traditional Endotracheal Tube
Number analyzed (Participants) | 30 | 30
Participants
  The overall incidence of displacement | 0 | 22
  Mild displacement | 0 | 11
  Moderate displacement | 0 | 8
  Severe displacement | 0 | 3
Statistical Analysis 1: Comparison: Prone Ventilation Endotracheal Tube vs the Traditional Endotracheal Tube; Test type: Superiority or Other; p < 0.05, Chi-squared; Odds Ratio (OR) = 0.73

2. Secondary Outcome: The Number of the Prolapse of Endotracheal Tube
Description: Counting the number who occured the prolapse of endotracheal tube in both groups
Time Frame: At any time within the procedure of the whole surgery
Population: All participants in both groups were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Prone Ventilation Endotracheal Tube | the Traditional Endotracheal Tube
Number analyzed (Participants) | 30 | 30
Participants | 0 | 0
Statistical Analysis 1: Comparison: Prone Ventilation Endotracheal Tube vs the Traditional Endotracheal Tube; Test type: Superiority or Other; p > 0.05, Chi-squared

3. Secondary Outcome: the Degree of Loose or Dampness of the Tape
Description: counting and quantifying the number who occured the dampness or loose of the tape in both groups
Time Frame: at the time when patients were turning to supine position
Population: all participants in both groups were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | the Traditional Endotracheal Tube | Prone Ventilation Endotracheal Tube
Number analyzed (Participants) | 30 | 30
Participants | 7 | 0

4. Other Pre Specified Outcome: the Incidence of Dysphagia
Description: count the number who suffered the dysphagia within the first 24 hours after extubation
Time Frame: within the first 24 hours after extubation
Population: all patients were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | the Traditional Endotracheal Tube | Prone Ventilation Endotracheal Tube
Number analyzed (Participants) | 30 | 30
Participants | 0 | 0

5. Other Pre Specified Outcome: the Incidence of Sore Throat
Description: count the number who suffer sore throat within the first 24 hour after extubation
Time Frame: within the first 24 hour after extubation
Population: all patients in both groups were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | the Traditional Endotracheal Tube | Prone Ventilation Endotracheal Tube
Number analyzed (Participants) | 30 | 30
Participants | 1 | 1

6. Other Pre Specified Outcome: the Incidence of Dysphonia
Description: count the number who suffered dysphonia within the first 24 hour after extubation
Time Frame: within the first 24 hour after extubation
Population: all patients in both groups were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | the Traditional Endotracheal Tube | Prone Ventilation Endotracheal Tube
Number analyzed (Participants) | 30 | 30
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: within the postoperative 24 hours
Description: the incidence rate of sore throat, hoarseness, dysphagia in both groups at 24-hour follow-up has been collected and calculated.
Groups:
- Prone Position Endotracheal Tube; Traditional Endotracheal Tube: there was one patient in this group occuring mild sore throat,and none occured dysphagia, dysphonia.
Arm/Group | Prone Position Endotracheal Tube | Traditional Endotracheal Tube
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 1/30 | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prone Position Endotracheal Tube (N=30) | Traditional Endotracheal Tube (N=30)
Sore throat (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — after the extubation of endotracheal tube, we investigated the participates whether they occured the sore throat, and the severity.

LIMITATIONS AND CAVEATS:
No limitations and caveats.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes